CLINICAL TRIAL: NCT00943865
Title: Effect of Three Lifestyle Interventions on Endothelial Function, Anthropometric Parameters and Cardiometabolic Profile in Obese Patients With Metabolic Syndrome: a Randomized Controlled Trial .
Brief Title: Three Lifestyle Interventions on Endothelial Function and Cardiometabolic Risk in Obese Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Beatriz Graeff Santos Seligman/ professor Serviço de Medicina Interna, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07033; GPPG07033 HCPA FIPE
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: metabolic syndrome; lifestyle; exercise; endothelial dysfunction; insulin sensitivity; lipids
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Motor Activity; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- hypocaloric diet + exercise advice (Active Comparator): Group 1 (control: tailored hypocaloric diet and exercise advised): patients received individually tailored hypocaloric diet, with 20% of total calories as fat (with 7-8 % of saturated fats), 50 to 65% carbohydrates and 15% to 20% proteins. Total of calories for each patient calculated assuming the ideal body weight to fulfill a BMI of 25 kg⁄ M2. Total daily amount of calories estimated calculating 30 calories/Kg of ideal weight for each subject. Subjects were advised against consuming high fat snacks or additional fats. Alimentary plans specified the number of servings from each food group, and dairy intake was held constant. Exercise was advised but not measured: they received recommendations to be physically active and perform 1 hour of aerobic exercise as preferred, everyday.
  Interventions: Behavioral: hypocaloric diet; Behavioral: Exercise recommendations
- pragmatic diet+ pedometer 10000 steps (Experimental): Group 2 (pragmatic diet + step counter) - Patients received a portable colored handbook with evidence- based recommendations on healthy eating attitudes and pragmatic menus, with low carbohydrates and high protein and vegetables. It included controlled portions (adjusted for individual hand size) for the six meals, with low glucose aliments and whole grains, legumes, yogurt, fruits, olive oils, eggwhite and low fat milk, fiber and a handful of nuts. Portions were tailored according to individual hand size, without calories counting. Beans, farofa and white cheese bread, which are commonly present in Brazilian food, and red meat were allowed, but with portion control. Subjects were provided with pedometers and were instructed to perform at least 10.000 steps daily, diary recorded.
  Interventions: Behavioral: Pragmatic diet; Behavioral: Pedometer-based fitness (10,000 steps)
- pragmatic diet + fitness (Experimental): Group 3 (pragmatic diet + fitness) - They received the same diet intervention (low carbohydrates, high protein and vegetables style diet and favoring daily brazilian cook habits colored handbook) and hand sized portion control instructions of group 2. They were scheduled for a more structured assisted exercise intervention: three bicycle ergometer sessions per week, under direct supervision of the same trained exercise physiologists in each session. Heart rate monitors were used to adjust workload to achieve the target heart rate (75% of the maximum attainable heart rate), as determined by their individual maximal treadmill exercise test. All patients were trained by the same staff, Borg scale was registered in every session and persuasive goal setting was made during exercise sessions.
  Interventions: Behavioral: Pragmatic diet; Behavioral: Structured assisted exercise (fitness)

INTERVENTIONS:
Behavioral: hypocaloric diet — patients received individually tailored hypocaloric diet, with 20% of total calories as fat (with 7-8 % of saturated fats), 50 to 65% carbohydrates and 15% to 20% proteins. Total of calories for each patient calculated assuming the ideal body weight to fulfill a BMI of 25 kg⁄ M2. Total daily amount of calories estimated calculating 30 calories/Kg of ideal weight for each subject. Subjects were advised against consuming high fat snacks or additional fats. Alimentary plans specified the number of servings from each food group, and dairy intake was held constant.
  Arms: hypocaloric diet + exercise advice
Behavioral: Exercise recommendations — Exercise was advised but not measured: they received recommendations to be physically active and perform 1 hour of aerobic exercise as preferred, everyday.
  Arms: hypocaloric diet + exercise advice
Behavioral: Pragmatic diet — Patients received a portable colored handbook with evidence- based recommendations on healthy eating attitudes and pragmatic menus, with low carbohydrates and high protein and vegetables. It included controlled portions (adjusted for individual hand size) for the six meals, with low glucose aliments and whole grains, legumes, yogurt, fruits, olive oils, eggwhite and low fat milk, fiber and a handful of nuts. Portions were tailored according to individual hand size, without calories counting. Beans, farofa and white cheese bread, which are commonly present in Brazilian food, and red meat were allowed, but with portion control.
  Arms: pragmatic diet + fitness; pragmatic diet+ pedometer 10000 steps
Behavioral: Pedometer-based fitness (10,000 steps) — Subjects were provided with pedometers and were instructed to perform at least 10,000 steps daily, diary recorded.
  Arms: pragmatic diet+ pedometer 10000 steps
Behavioral: Structured assisted exercise (fitness) — They were scheduled for a more structured assisted exercise intervention: three bicycle ergometer sessions per week, under direct supervision of the same trained exercise physiologists in each session. Heart rate monitors were used to adjust workload to achieve the target heart rate (75% of the maximum attainable heart rate), as determined by their individual maximal treadmill exercise test. All patients were trained by the same staff, Borg scale was registered in every session and persuasive goal setting was made during exercise sessions
  Arms: pragmatic diet + fitness

SUMMARY:
Obese patients with metabolic syndrome without diabetes or ischemic heart disease were randomized to three lifestyle interventions: 1. hypocaloric tailored diet with standard recommendations 2. pragmatic healthy style diet adapted to brazilian habits with portion control and pedometers to perform 10000 steps daily recorded or 3. pragmatic healthy style diet adapted to brazilian habits with portion control plus fitness three times a week under direct supervision. The main outcome was brachial reactivity, a surrogate marker of atherosclerosis, and secondary outcomes were cardiometabolic profile, arterial pressure and anthropometric measures: weight,waist circumference and bioimpedanciometry to access fat proportion and insulin sensitivity.

DETAILED DESCRIPTION:
It's a 12 week single center randomized controlled trial to evaluate three different lifestyle interventions on flow mediated vasodilatation, cardiometabolic profile and anthropometric parameters in non-diabetic persons with metabolic syndrome without coronary heart disease.

After informed consent, they will be randomized to 3 different lifestyle interventions: 1. Hypocaloric tailored AHA type 1 diet plus standard exercise advice; 2. Pragmatic portion controlled healthy diet plus pedometers to perform 10.000 steps daily or 3. pragmatic portion controlled healthy diet plus fitness under direct supervision,using heart rate monitors to adjust workload to achieve the target heart rate (75% of the maximum attainable heart rate - HRpeak, as determined by their individual maximal treadmill exercise test).Main outcome is endothelium vasodilation accessed through brachial ultrasound, a surrogate marker of atherosclerosis. Secondary outcomes are anthropometric data: weight, waist circumference and fat proportion, cardiometabolic profile and insulin sensitivity (HOMA-R).

ELIGIBILITY:
Inclusion Criteria:

* men and women 30-55 years with BMI 30-40 and waist 95 cm or more
* normal OGTT
* normal treadmill stress test
* plus 2 of 4:

  1. low serum levels of HDL cholesterol (<40 mg⁄dL for men or < 50 mg ⁄dL for women);
  2. hypertriglyceridemia (triglyceride levels of 150 mg⁄dL or greater);
  3. impaired glucose homeostasis (fasting plasma glucose concentration of 110 mg⁄dL or greater or glucose of 140 mg⁄dL or greater after OGTT or
  4. hypertension (systolic blood pressure ≥ 140 or diastolic blood pressure ≥90 mmHg or treatment with antihypertensive drugs).

Exclusion Criteria:

* diabetes
* ischemic heart disease or any abnormality on treadmill stress test
* inflammatory or chronic disorder
* pregnancy
* lactation
* creatinine level of 1,5 mg/dL or more
* gastrointestinal problems or musculoskeletal disorders that would prevent them to follow the test diets or exercise interventions
* liver dysfunction with a factor of at least 3 above the upper limit of normal in AST and ALT levels
* thyroid dysfunction, with serum TSH out of normal limits
* use of immunosuppressive drugs, corticosteroids or anorexigen

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
endothelial mediated vasodilation | at enrollment, after 6 and after 12 weeks

SECONDARY OUTCOMES:
weight | randomization, 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz G Seligman, MD MsC, Principal Investigator — Serviço de Medicina Interna Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil